CLINICAL TRIAL: NCT02301780
Title: Combined Multi-marker Screening and Randomised Patient Treatment With Aspirin for Evidence-based Pre-eclampsia Prevention. University College London - Sponsor of All EU Study Sites.
Brief Title: Combined Multi-marker Screening and Treatment With Aspirin for Pre-eclampsia Prevention
Acronym: ASPRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0066-14-RMC
Record Dates: First submitted 2014-11-23; First posted 2014-11-26 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Intervention Group (Active Comparator): Aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Participants who are screened with a high-risk of developing PET will be randomised into one of 2 arms of the trial (on the same day as screening or within 1 week of the screening visit). Randomised participants will be advised to start 150mg of Aspirin/Placebo once per night within 24 hours of randomisation until 36 weeks' gestation or when signs of labour commence.
  The maximum duration for aspirin or placebo intake will be 180 days.
  Arms: Intervention Group
Drug: Placebo — Participants who are screened with a high-risk of developing PET will be randomised into one of 2 arms of the trial (on the same day as screening or within 1 week of the screening visit). Randomised participants will be advised to start 150mg of Aspirin/Placebo once per night within 24 hours of randomisation until 36 weeks' gestation or when signs of labour commence.
  The maximum duration for aspirin or placebo intake will be 180 days.
  Other Names: Aspirin
  Arms: Control Group

SUMMARY:
Phase III two arm double-blinded randomised controlled trial to examine the effect of prophylactic low-dose aspirin from the first-trimester of pregnancy in women at increased risk for PET on the incidence and severity of the disease

DETAILED DESCRIPTION:
Screening and Prevention of Pre-eclampsia (High Blood Pressure): Randomised Trial of Aspirin Versus Placebo (ASPRE)

Screening: All women with singleton pregnancies undergoing routine screening for aneuploidies will be invited to participate in the screening study for PET.

Interventions: Participants who are screened with a high-risk of developing PET will be randomised into one of 2 arms of the trial (on the same day as screening or within 1 week of the screening visit). Randomised participants will be advised to start 150mg of Aspirin/Placebo once per night within 24 hours of randomisation until 36 weeks' gestation or when signs of labour commence.

The maximum duration for aspirin or placebo intake will be 180 days.

Key Inclusion and Exclusion Criteria Inclusion criteria for participant selection for RCT Age > 18 years, Singleton pregnancies, Live fetus at 11-13 weeks of gestation, High-risk for preterm-PET at 11-13 weeks by the algorithm combining maternal history and characteristics, biophysical findings (mean arterial pressure and uterine artery Dopplers) and biochemical factors (pregnancy associated plasma protein-A and placental growth factor), English, Italian, Spanish, French, Dutch or Greek speaking (otherwise interpreters will be used), Informed and written consent.

Exclusion criteria Multiple pregnancies, Women taking low-dose aspirin regularly (administration must have ceased >28days prior to randomisation), Pregnancies complicated by major fetal abnormality identified at the 11-13 weeks assessment, Women who are unconscious or severely ill, those with learning difficulties, or serious mental illness, Bleeding disorders such as Von Willebrand's disease, Peptic ulceration, Hypersensitivity to aspirin or already on long term non-steroidal anti-inflammatory medication, Age < 18 years, Concurrent participation in another drug trial or at any time within the previous 28 days, Any other reason the clinical investigators think will prevent the potential participant from complying with the trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Singleton pregnancies
* Live fetus at 11-13 weeks of gestation,
* High-risk for preterm-PET at 11-13 weeks by the algorithm combining maternal history and characteristics, biophysical findings (mean arterial pressure and uterine artery Dopplers) and biochemical factors (pregnancy associated plasma protein-A and placental growth factor),
* English, Italian, Spanish, French, Flemish, Hebrew, Arabic and Russian speaking (otherwise interpreters will be used)
* Informed and written consent.

Exclusion Criteria:

* Multiple pregnancies
* Women taking low-dose aspirin regularly
* Pregnancies complicated by major fetal abnormality identified at the 11-13 weeks assessment
* Women who are unconscious or severely ill, those with learning difficulties, or serious mental illness, Bleeding disorders such as Von Willebrand's disease
* Peptic ulceration
* Hypersensitivity to aspirin or already on long term nonsteroidal anti- inflammatory medication
* Age < 18 years
* Concurrent participation in another drug trial or at any time within the previous 28 days
* Any other reason the clinical investigators think will prevent the potential participant from complying with the trial protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Pre-eclampsia requiring delivery prior to 37 weeks of gestation | 24-26 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No